CLINICAL TRIAL: NCT01506258
Title: Effects of the Infusion of Autologous Non-cryopreserved CD34+ Cells in Newborns With Asphyxia
Brief Title: Autologous Stem Cells in Newborns With Oxygen Deprivation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Consuelo Mancias Guerra, Pediatric Hematology Professor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-11-011
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Apgar; 0-3 at 1 Minute; Metabolic Acidosis; Hypoxia, Brain; Multiple Organ Failure
Keywords: CD34+; perinatal hypoxia; autologous hematopoietic stem cells; cord and placental blood; cerebral palsy
MeSH Terms: conditions — Acidosis; Hypoxia, Brain; Multiple Organ Failure; Cone-Rod Dystrophies; Cerebral Palsy | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients not infused with stem cells (No Intervention): Historic Controls
  Interventions: Procedure: Observation
- Patients infused with stem cells (Experimental)
  Interventions: Procedure: Application of Stem Cells

INTERVENTIONS:
Procedure: Application of Stem Cells — IV infusion of autologous stem cells within the first 48 hours after birth.
  Other Names: IV infusion of autologous cord and placental cord blood
  Arms: Patients infused with stem cells
Procedure: Observation — Control group of patients that meet the inclusion criteria but that do not wish to have the intervention.
  Other Names: Comparison group
  Arms: Patients not infused with stem cells

SUMMARY:
The purpose of this study is to determine whether the plasticity of autologous intravenous application of cord blood stem cells would improve the clinical course of asphyxiated newborns.

DETAILED DESCRIPTION:
When there is oxygen deprivation, more frequently in premature newborns, the brain and other organs suffer severe consequences. There is evidence that hematopoietic stem cells can help in this scenario by promoting the release of growth-enhancing factors that can help control the damage due to their "homing" capacity, which attracts them to injured sites.

Cord and placental blood have a high concentration of these stem cells, and because its obtention is relatively easy, it seems like a feasible treatment in perinatal hypoxia.

There are current clinical trials that use cryopreserved cord blood for these patients but, to do that, the stem cells have to be frozen and then thawed to be infused, losing a considerable amount of stem cells (almost half of them). We want to evaluate the same condition but infusing non-cryopreserved autologous cord and placental blood because we believe it can be more beneficial due to the greater amount of cells infused, the avoidance of the cryoprotection agent´s toxicity and the lower costs.

ELIGIBILITY:
Inclusion Criteria:

* Apgar < 5 at 5 minutes
* Mixed or metabolic acidosis with a pH <7.0 from umbilical cord blood sample
* Neurological manifestations compatible with Hypoxic-Ischemic Encephalopathy
* Any degree of organic/systemic affectation (cardiovascular, gastrointestinal, hematologic and/or respiratory)

Exclusion Criteria:

* Neurodegenerative, autoimmune or genetic disease
* Active infection at birth
* Informed Consent not signed

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Effects of Stem Cell Infusion at 1 week after discharge | 1 week
  Clinical assessment, including the Amiel-Tison Neurological Assessment
Effects of Stem Cell Infusion at 1 year after discharge | 1 year
  Clinical assessment, including the Amiel-Tison Neurological Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo Mancias-Guerra, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez; Alma R Marroquin-Escamilla, MD, Study Director — Hospital Universitario Dr. Jose E. Gonzalez; David Gómez-Almaguer, MD, Study Chair — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Neonatology Department of the Pediatrics Service, Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico